CLINICAL TRIAL: NCT06077357
Title: Evaluation of Frailty, Hand Grip Strength, Physically Activity, Kinesiophobia and Fatigue in Chronic Obstructive Pulmonary Disease and Asymptomatic Geriatric Individual
Brief Title: Evaluation in Individuals with COPD and Asymptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meral SERTEL, ASSOCIATE PROFESSOR DOCTOR, Kırıkkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KU-FTR-IK-01
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pain; Muscle Strength; Kinesiophobia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Two groups consisting of a COPD group and an Asymptomatic group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD Patients (Active Comparator): Having COPD. Older than 65 years old and not having any communication problems.
  Interventions: Other: MMSE Test; Other: PASE Test; Other: The PRISMA-7 Frailty Scale; Other: TAMPA Test; Other: (JAMAR) Muscle Test; Other: Fatigue Severity Scale
- Asymptomatic Patients (Active Comparator): Not having a diagnosis of COPD and being over 65 years old and not having any communication problems.
  Interventions: Other: MMSE Test; Other: PASE Test; Other: The PRISMA-7 Frailty Scale; Other: TAMPA Test; Other: (JAMAR) Muscle Test; Other: Fatigue Severity Scale

INTERVENTIONS:
Other: MMSE Test — Mini Mental State Examination (MMSE), is a brief mental test used to assess individuals' cognitive functions. This test evaluates basic cognitive abilities such as memory, attention, calculation, language, orientation, and problem-solving. MMSE is commonly used for monitoring and assessing mild cognitive impairments, dementia, and other neurological conditions. This test is typically scored out of 30, with higher scores indicating better cognitive function.
Other: PASE Test — The PASE test stands for "Physical Activity Scale for the Elderly." This scale is used to assess the physical activities undertaken by elderly individuals in their daily lives. The PASE test allows for the evaluation of both daily activities such as walking, climbing stairs, and household chores, as well as exercise routines. It is used to determine the level of physical activity in elderly individuals and support the process of healthy aging.
Other: The PRISMA-7 Frailty Scale — The PRISMA-7 Frailty Scale is a tool used to assess the level of frailty in elderly individuals. This scale evaluates signs of frailty such as physical activity, fatigue, weight loss, and difficulties with vision and hearing. PRISMA-7 is employed in determining the risk of frailty in the elderly and aids in identifying appropriate treatment and support methods.
Other: TAMPA Test — The TAMPA test, abbreviated from "Tampa Scale for Kinesiophobia," is a scale used to assess fears related to pain. This scale is employed to evaluate the fear of pain and avoidance behaviors associated with it. By measuring individuals' attitudes and fears towards pain, the TAMPA test helps identify their emotional and behavioral responses in this area.
Other: (JAMAR) Muscle Test — The JAMAR Muscle Test is a widely used clinical assessment tool for evaluating hand grip strength. It involves using a device called a dynamometer to measure the force exerted by a person's hand when squeezing the instrument. This test provides valuable information about an individual's upper body strength, which can be important in various medical and rehabilitative contexts. The JAMAR Muscle Test is often utilized in physical therapy, sports medicine, and other healthcare fields.
Other: Fatigue Severity Scale — The Fatigue Severity Scale (FSS) is a self-report questionnaire used to assess the severity of fatigue in individuals. It consists of nine items that measure the impact of fatigue on various aspects of daily life, such as physical functioning, motivation, and mental clarity. The FSS is commonly used in clinical settings and research studies to quantify the level of fatigue experienced by individuals with various medical conditions, including chronic illnesses, neurological disorders, and mental health conditions. It provides valuable information for healthcare professionals in understanding and managing fatigue-related symptoms.

SUMMARY:
The literature does not provide sufficient information on the evaluation of frailty, handgrip strength, physical activity, kinesiophobia, and fatigue in elderly individuals with Chronic Obstructive Pulmonary Disease and asymptomatic elderly individuals. Additionally, there is a gap in the literature regarding the impact of COPD on these parameters in geriatric individuals diagnosed with Chronic Obstructive Pulmonary Disease . To fill this gap in the literature and to establish treatment approaches based on the results of parameters studied in elderly individuals with Chronic Obstructive Pulmonary Disease in future studies.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a prevalent condition among the elderly population, considered a leading cause of morbidity and mortality. It is characterized by chronic inflammatory responses associated with harmful particles or gases in the airways and lungs, resulting in persistent airflow limitation that is both preventable and treatable . While cough and sputum are reported as clinical symptoms in COPD cases, the most prominent clinical symptom is dyspnea. Age-related physiological changes and frailty lead to a decrease in levels of physical activity. The resulting deconditioning from reduced physical activity causes a decline in ventilation quality, creating a vicious cycle that progressively exacerbates dyspnea. This study involves the comparison of individuals diagnosed with COPD with asymptomatic geriatric individuals. Its aim is to examine the effects of COPD on frailty, handgrip strength, physical activity, kinesiophobia, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for COPD Patients:

  * Having received a diagnosis of COPD
  * Being 65 years of age or older
  * Volunteering to participate in the study
  * Not having any mental or communication issues that would hinder the completion of the questionnaires to be used in the research
* Inclusion Criteria for Asymptomatic Individuals:

  * Not having received a diagnosis of COPD
  * Being 65 years of age or older
  * Volunteering to participate in the study
  * Not having any mental or communication issues that would hinder the completion of the questionnaires to be used in the research

Exclusion Criteria:

* Exclusion Criteria for COPD and Asymptomatic Individuals:

  * Having a diagnosis of both physical and mental illnesses
  * Being diagnosed with unstable COPD
  * Having conditions such as unstable angina, prior heart attack, uncontrolled hypertension, cancer, and neurological disorders accompanied by functional limitations
  * Currently being addicted to alcohol or substances
  * Having severe visual and hearing impairments
  * Having undergone major surgery in the past few months
  * Having a history of recurring significant clinical infections.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
The Fatigue Severity Scale | 4 months
  The Fatigue Severity Scale evaluates the severity of fatigue through 9 questions, with scores ranging from 9 to 63 on the scale. Each question is scored on a 1 (completely disagree) to 7 (completely agree) Likert scale. A higher score indicates increased severity of fatigue.A higher score is worse.

SECONDARY OUTCOMES:
The Physical Activity Scale for the Elderly (PASE) | 4 months
  The questionnaire assesses the physical activities of elderly individuals within the past week, covering components related to leisure, household chores, and work-related physical activities. Participation in leisure-time activities, including outdoor walking of light, moderate, and vigorous intensity, as well as muscle-strengthening exercises, is recorded as never, seldom (1-2 days/week), sometimes (3-4 days/week), and often (5-7 days/week). Additionally, the duration of activities is classified as less than 1 hour, 1-2 hours, 2-4 hours, and more than 4 hours. A higher score indicates higher physical activity levels.A higher score is better.
The Tampa Scale of Kinesiophobia | 4 months
  The Tampa Scale of Kinesiophobia is a 17-item checklist. A 4-point scale is used for scoring (1= Strongly Disagree, 4= Strongly Agree). Individuals receive a total score between 17 and 68. A higher score indicates higher levels of kinesiophobia.A higher score is worse.
Hand Grip Strength Measurement | 4 months
  Hand Grip Strength Measurement is a test used to assess upper extremity muscle strength. The test is performed three times on both hands, and the results are recorded. The highest values on both sides are documented. A high score indicates high hand grip strength.
PRISMA-7 Fragility Test | 4 months
  This scale consists of 7 questions. Each question is answered with yes or no. Having more "yes" answers indicates a higher level of frailty. Having 3 or more "yes" answers indicates fragility.A higher score is worse.
The Mini Mental Test (MMT) | 4 months
  This test is conducted for cognitive assessment. Scores range from 0 to 30. A score higher than 24 indicates no cognitive impairment.A higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Meral SERTEL, Doc.Dr., Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale Yuksek Ihtisas Hospital, Kırıkkale, Yahsihan, Turkey (Türkiye)